CLINICAL TRIAL: NCT05992857
Title: Randomized Controlled Trial Comparing Pancreaticoduodenectomies With or Without Complete Arterial Coverage by Omentoplasty in Patients With High Risk of Postoperative Pancreatic Fistula.
Brief Title: Pancreaticoduodenectomies With Complete Arterial Coverage by Retromesenteric Omentoplasty
Acronym: PACOMARCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220823
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pancreatectomy; Complication of Surgical Procedure
Keywords: Pancreaticoduodenectomy; Post-pancreatectomy haemorrhage; Omentoplasty; Post-operative pancreatic fistula
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Intervention Model Description: National, Phase IIIb multicenter, centrally randomized open-label trial with two parallel arms. Participants will be distributed between the two arms at a ratio (1:1).
  Randomization will be built by block of unequal size stratified by center and the prophylactic use of somatostatin/octreotide-Yes/No
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retromesenteric omental flap covering all exposed peripancreatic arteries (Experimental): A J-shaped omental flap is created by extensive mobilization of the greater omentum, and if needed, lengthening by division of vertical collaterals of gastroepiploic vessels section or thinning it out in patients with visceral obesity. This omental flap is ascended through the retromesentric route to cover all the peri-pancreatic vessels at risk of bleeding after pancreatic resection (hepatic artery, proximal part of the splenic artery, superior mesenteric artery, and right hepatic artery originating from superior mesenteric artery when present)
  Interventions: Procedure: Pancreaticoduodenectomy with retromesenteric omental flap
- Control (Active Comparator): No omental flap or an omental flap not using the retromesenteric route and only interposed between the pancreatic anastomosis and the hepatic artery, or a single round ligament flap wrapping the hepatic artery only.
  Interventions: Procedure: Pancreaticoduodenectomy without retromesenteric omental flap

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy without retromesenteric omental flap — Resection of the pancreatic head, duodenum, distal common bile duct and gallbladder followed by reconstruction using pancreaticojejunostomy, hepaticojejunostomy, and gastrojejunostomy performed on the first jejunal loop.
  Arms: Control
Procedure: Pancreaticoduodenectomy with retromesenteric omental flap — All exposed peripancratic arteries should be covered with a retromesentric omental flap
  Arms: Retromesenteric omental flap covering all exposed peripancreatic arteries

SUMMARY:
To assess the efficacy of complete covering using retromesenteric omentoplasty vs. partial covering or no covering of peripancreatic arteries in decreasing incidence of grade B+C post-pancreatectomy hemorrhage (PPH), i.e. treated by transfusion and / or radiological or surgical hemostasis after PD in patients with high risk of POPF.

DETAILED DESCRIPTION:
Grade B+C postpancreatectomy hemorrhage (PPH) is a severe complication following pancreaticoduodenectomy (PD), more frequently observed in patients with high-risk of postoperative pancreatic fistula (POPF). To date no randomized controlled trial has assessed the impact of an omentoplasty covering all arteries exposed during PD on the prevention of clinically relevant postpancreatectomy hemorrhage (PPH) in patients with high-risk of POPF (fistula risk score between 7 to 10)

In the standard technique, no omental flap is used or an omental flap is only interposed between the pancreatic anastomosis and the hepatic artery, and/or the round ligament wraps the hepatic artery only. An orignal approach is proposed using a J-shaped omental flap created by the mobilization of the greater omentum and ascended through the retromesentric route to cover all the peri-pancreatic arteries at risk of bleeding after pancreatic resection.

Patient fulfilling eligibility criteria will be enrolled during a selection visit (V0) which may take place 45 days and up to 1 day prior PD surgery. Patient will be randomized intra-operatively either in the experimental arm or the control arm for allocation the omental covering technique.

After surgery, the following visits will be planned for the patient follow up:

* V2: End of hospitalization visit which can be done up to 1 day prior discharge.
* V3: POD 45 (±15) days which will take place at the hospital.
* Vai: Additional visit which may take place if the patient is readmitted for postoperative complication. Those visits may take place between V2 and V4 up to 1 day prior discharge.
* V4: POD 90 (±15) days is the end of study visit. It will take place at the hospital.

During those visits, data will be collected to validate the primary and secondary endpoints of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients requiring a pancreaticoduodenectomy (PD) for any indication
* Open approach
* Affiliation to the French public healthcare insurance
* Fistula risk score (FRS) ≥ 7 confirmed intraoperatively
* Ability to understand and to comply with the study protocol
* Reconstruction with PJ and external pancreatic stent
* Signed written informed consent
* Inclusion is allowed for patients:

  * On curative or long-term anticoagulation or aspirin (indicated for previous thromboembolic complications, heart disease, previous history of stroke)
  * Undergoing PD with venous resection

Exclusion Criteria:

* Presence of distant tumor deposits (liver and peritoneal metastases, and/or para-aortic lymph nodes metastases) reveals during intraoperative exploration for patient with malignant pancreatic or periampullary tumor.
* Patients with previous abdominal surgery compromising completion of retromesenteric omentoplasty
* PD with arterial resection (i.e. resection of hepatic artery, splenic artery, superior mesenteric artery, or celiac axis)
* Laparoscopic or robotic PD
* Reconstruction wih pancreatico-gastrostomy
* Total pancreatectomy
* Emergency procedure
* Pregnant women
* Patient under guardianship and curatorship
* Participation in another interventional study evaluating complication after pancreaticoduodenectomy or patient still being in the exclusion period at the end of a previous study evaluating drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of postpancreatectomy haemorrhage clinically significant (graded B or C) | From surgery to post-operative day 90
  According to the definition of the International Study Group of Pancreatic Surgery (ISGPS)
  * Grade B: PPH is early (< 24h) or late bleeding without any organ failure
  * Grade C: PPH is late bleeding with organ failure (hemodynamic, renal, cardiac, respiratory failure)
  * Both grade B and C bleeding require transfusion and/or a procedure to obtain hemostasis including radiological embolization, endoscopic intervention or reoperation.

SECONDARY OUTCOMES:
Mortality | From surgery to post-operative day 90
Overall Morbidity | From surgery to post-operative day 90
  Assessed by comprehensive complication index (CCI)
Rate of grade B+C post-operative pancreatic fistula | From post-operative day 3 to post-operative day 90
  According to 2016 ISGPF classification (Bassi C et al. 2016) :
  -Amylase level in the drainage fluid (or fluid of any collection) exceeding 3 times the upper limit of local laboratory norm of serum amylase level co-existing with clinically significant deviation from the normal post operative course.
Rate of grade A post-pancreatectomy haemorrhage | From surgery to post-operative day 90
  [12:51] Alain (Invité)
  Post pancreatectomy haemorrhage requiring neither transfusion nor hemostatic procedure
Hospital readmission | From end of initial hospital stay to post-operative day 90
  Defined by unplanned readmission
Total duration of hospital stay | From surgery to post-operative day 90
  Including duration of initial stay and readmision if present
Rate of arterial pseudoaneurysm | Performed at post-operative day 90
  Detected by routine enhanced CT with intravenous contrast injection

CONTACTS AND LOCATIONS:
Overall Officials: Alain SAUVANET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Beaujon Hospital, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided